CLINICAL TRIAL: NCT02472509
Title: The Role of Ursodeoxycholic Acid in Treatment of Gallstones in Hemolytic Disorders
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study not feasible - very low recruitment rate
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Ursolit_Hemolytic disorders
Record Dates: First submitted 2015-02-04; First posted 2015-06-16 (Estimated); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Hemolytic Disorders; Gallstones
Keywords: Ursodeoxycholic acid (UDCA); White blood cells (WBC); Alanine Transaminase (ALT); Alkaline Phosphatase (ALP); Aspartate Aminotransferase (AST); Gamma-Glutamyl Transpeptidase (GGT); Lactate dehydrogenase (LDH); Low-Density Lipoprotein (LDL); High-Density Lipoprotein (HDL); Glucose-6-phosphate dehydrogenase (G6PD); Ultrasound (US)
MeSH Terms: conditions — Gallstones | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open Label (Experimental): 32 patients with hemolytic disorders meeting the inclusion and exclusion criteria will be commenced on Ursodeoxycholic acid (UDCA).
  Interventions: Drug: Ursodeoxycholic Acid

INTERVENTIONS:
Drug: Ursodeoxycholic Acid — Patients will be commenced on UDCA 15mg/kg/day (maximum dose 900mg/day) in 2-3 divided doses for 12 months.
  Patients who are unable to tolerate tablet medication will be started on UDCA syrup at the same dose.
  Other Names: Ursolit

SUMMARY:
It is well established that hemolytic diseases predispose patients to the development of pigment gallstones. Gallstones are noted in at least 5% of children under the age of 10 years, increasing to 40-50% in the second to fifth decades. The co-inheritance of Gilbert's syndrome increases the risk of cholelithiasis four to five-fold.

In patients with chronic hemolysis, total bile lipid concentration is decreased and the total bilirubin to total lipid ratio is increased. This suggests that the conjugating capacity of hepatocytes is surpassed by the excessive amount of bilirubin resulting from hemolysis. Increased bilirubin monoconjugate and unconjugated bilirubin can precipitate in bile and form complexes with inorganic ions, mostly calcium, and develop into stones.

Patients with hemolytic disorders can also develop biliary sludge, a suspension of precipitated particulate matter in bile dispersed in a viscous, mucin-rich liquid phase . The chemical composition of the precipitates correlates well with the composition of the associated stone and sludge often stands as a harbinger of future stone development.

There is strong data suggesting a benefit in treating cholelithiasis with UDCA and also in preventing gallstone development in various high risk scenarios.

There are several proposed mechanisms for the positive effect of UDCA in primary prevention of pigment stones. Mucoglycoproteins are present in significant amounts in black pigment stones and contribute to the matrix of gallstones. UDCA suppresses the secretion of protein and decreases the levels of various proteins in bile . It has also been suggested that increased colonic bile salt may solubilize unconjugated bilirubin and may prevent calcium complexing.

There is no published data at present on the role of UDCA in prevention and treatment of cholelithiasis in hemolytic diseases. The investigators hypothesise that UDCA can be of benefit to patients with hemolytic disorders in the primary prevention of pigment stones, possible resolution of biliary sludge and existent stones, and reduction of symptomatic episodes of cholelithiasis.

DETAILED DESCRIPTION:
The research protocol extends for up to 12 months, during which the participant will attend 3 clinic visits at Shaare Zedek Medical Centre; one at study enrollment, one at 6 months and one at 12 months.

All patients identified will have their medical records reviewed for previous clinical, biochemical or sonographic evidence of gallstones.

Patients will undergo a baseline abdominal ultrasound to assess for biliary sludge, gallstones, or evidence of previous cholecystitis (eg. Thickened gallbladder wall).

All patients will also have blood tested for liver biochemistry, complete blood count, hemolytic screen and fasting lipids.

Participants will be commenced on UDCA 15mg/kg/day (maximum dose 900mg/day) in 2-3 divided doses for 12 months.

Patients who are unable to tolerate tablet medication will be started on UDCA syrup at the same dose.

Each of the in-house visits will include:

1. An explicit history taking and review of patient's notes, including review of symptoms, blood tests and previous ultrasounds, other medical conditions and medications.
2. Physical examination - including measuring splenic size, assessing for right upper quadrant abdominal tenderness
3. Blood tests

   1. Hemoglobin, WBC
   2. Liver biochemistry: ALT, AST, GGT, ALP (Alkaline Phosphatase), Bilirubin (conjugated and unconjugated), Albumin
   3. Hemolytic screen: LDH, haptoglobin, reticulocytes
   4. Fasting lipids: LDL, HDL, Triglycerides

Repeat abdominal ultrasound will be performed at 12 months. The US will specifically relate to the following features in comparison to the baseline US:

1. Presence of biliary sludge
2. Presence of gallstone: i.Size ii.Number
3. Presence of bile duct dilatation
4. Presence of gall bladder wall thickening

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of a hemolytic disorder including spherocytosis, G6PD deficiency, thalassemia or sickle cell disease.
2. Patients with cholelithiasis or bile sludge.
3. Age greater than or equal to 4 years.
4. Ability to consent to and participate in the study and follow study procedures.

Exclusion Criteria:

1. Previous splenectomy (complete or partial)
2. Evidence of hemolytic crisis at the time of research enrollment
3. Patients with highly symptomatic gallstones who have planned surgical intervention
4. Known allergy or intolerance to UDCA
5. Existence of concurrent hepatic disease
6. Any other laboratory or clinical condition that the investigator considers clinically significant that could impact the outcome of the study or the safety of the patient.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-12; Primary Completion 2017-09-10 (Actual); Study Completion 2017-09-10 (Actual)

PRIMARY OUTCOMES:
Lack of sonographic, clinical or biochemical evidence of progression of cholelithiasis or biliary sludge. | 12 months

SECONDARY OUTCOMES:
Improvement in number and severity of episodes of symptomatic gallstones. | 12 months
Rate of surgical intervention for gallstones disease. | 12 months
Sonographic improvement (size and number of gallstones, presence of bile sludge, gallbladder wall thickness). | 12 months
Evaluate tolerability and adverse effects of UDCA therapy in hemolytic disorders. | 12 months
  including non-specific abdominal discomfort, rash or nausea.
Improved biochemical evidence of gallstone disease | 12m
  reduced gamma-glutamyl-transpeptidase (GGT) and alkaline phosphatase (ALP).

CONTACTS AND LOCATIONS:
Overall Officials: Oren Ledder, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel